CLINICAL TRIAL: NCT05440383
Title: A Phase III Confirmatory Study of KLH-2109 in Uterine Fibroids Patient With Menorrhagia
Brief Title: A Clinical Study of KLH-2109 in Uterine Fibroids Patient With Menorrhagia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KLH2301
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Uterine Fibroids (MeSH Heading: Leiomyoma)
MeSH Terms: conditions — Leiomyoma | interventions — linzagolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KLH-2109 (Experimental): Oral administration
  Interventions: Drug: KLH-2109
- Leuprorelin (Active Comparator): Subcutaneous administration
  Interventions: Drug: Leuprorelin

INTERVENTIONS:
Drug: KLH-2109 — Oral administration
  Arms: KLH-2109
Drug: Leuprorelin — Subcutaneous administration
  Arms: Leuprorelin

SUMMARY:
Multi-center, randomized, double-blind, parallel-group study to confirm non-inferiority of KLH-2109 to Leuprorelin acetate in uterine fibroids patient with menorrhagia

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Japanese woman diagnosed with uterine fibroids
* Patients confirmed by transvaginal ultrasonography to have at least 1 myoma that meet all of the following conditions:
* Larger than a certain standard
* No calcification
* Not receiving surgical treatment
* Patients with a normal menstrual cycle
* Patients diagnosed with menorrhagia

Exclusion Criteria:

* Patients with complication or history of blood system diseases (salasemia, sickle erythrocyte anemia, folic acid deficiency, coagulation disorder, etc.) (excluding iron deficiency anemia and latent iron deficiency anemia)
* Patients with lower abdominal pain due to irritable bowel syndrome or lower abdominal pain due to severe interstitial cystitis
* Patients with undiagnosed abnormal genital bleeding

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a total PBAC score of less than 10 from Week 6 to 12 after beginning of study drug administration | Up to 12 weeks
  PBAC (pictorial blood loss assessment chart) score

SECONDARY OUTCOMES:
Proportion of subjects with a total PBAC score of less than 10 from Week 2 to 6 after beginning of study drug administration | Up to 24 weeks
  PBAC (pictorial blood loss assessment chart) score
Proportion of subjects with a total PBAC score of less than 10 from Week 18 to 24 after beginning of study drug administration | Up to 24 weeks
  PBAC (pictorial blood loss assessment chart) score
Proportion of subjects with a total PBAC score of less than 10 during 6 weeks before end of study drug administration | Up to 24 weeks
  PBAC (pictorial blood loss assessment chart) score
Change from baseline in blood hemoglobin | Up to 24 weeks
  Hemoglobin
Change rate from baseline in myoma volume | Up to 24 weeks
  Myoma volume
Change rate from baseline in uterine volume | Up to 24 weeks
  Uterine volume
Change from baseline in UFS-QOL score | Up to 24 weeks
  UFS-QOL (uterine fibroid symptom and QOL) score
Incidence of adverse events and adverse drug reactions | Up to 24 weeks
  Adverse events and adverse drug reactions
Change rate from baseline in bone metabolic markers (BAP and serum NTx) | Up to 24 weeks
  Bone metabolic markers (BAP and serum NTx)
Change rate from baseline in bone density (DXA) | Up to 24 weeks
  Bone density, T-score

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Clinical Resarch Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Undecided